CLINICAL TRIAL: NCT06603870
Title: Secondary Prevention of Venous Thromboembolism in Patients With Cancer and Catheter-Related Upper Extremity Deep Vein Thrombosis (STREAM-Line Study)
Brief Title: Secondary Prevention of VTE in Patients With Cancer and Catheter-Related Upper Extremity Deep Vein Thrombosis
Acronym: STREAM-Line
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STREAM-Line
Record Dates: First submitted 2024-07-16; First posted 2024-09-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism; Cancer; Upper Extremity Deep Vein Thrombosis; Catheter-Related Infections
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms; Upper Extremity Deep Vein Thrombosis; Catheter-Related Infections | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Apixaban 2.5 mg twice daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apixaban (Experimental): 2.5 mg twice daily
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban is Health Canada approved for routine treatment and secondary prevention of VTE. Upon enrollment and during follow-up, patients will be managed with a prophylactic dose of apixaban (2.5 mg orally twice daily) as long as either a CVC or active cancer is present. Apixaban will be stopped at the time of CVC removal and when cancer is in remission. Patients will be instructed to contact the study team when their CVC is removed (to determine if apixaban should be continued, based on cancer status at the time), or any thrombotic or bleeding concerns were to occur in between visits. The investigators will record loss to follow-up, drop out, or death during the study.

SUMMARY:
This trial seeks to evaluate a management strategy after the acute treatment duration (≥ 3 months of therapeutic anticoagulation) for patients with cancer and catheter-related upper extremity deep vein thrombosis (DVT).

DETAILED DESCRIPTION:
The aim of the STREAM-Line Trial is to demonstrate that the STREAM-Line management strategy is safe after the acute treatment duration (≥ 3 months of therapeutic anticoagulation) in patients with cancer and catheter-related upper extremity DVT. Upon enrollment and during follow-up, patients will be managed with a prophylactic dose of apixaban (2.5 mg orally twice daily) as long as either a central venous catheter (CVC) or active cancer is present (STREAM-Line management strategy). Apixaban will be stopped at the time of CVC removal and when cancer is in remission. Day 90±14 and Day 180+14 follow-up visit procedures will be done by phone call or in person.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) with active cancer, defined as cancer (other than localized non-melanoma skin cancer) diagnosed or treated within 6 months, or the presence of metastatic, recurrent, or progressive malignancy, ongoing anticancer therapy, or hematological malignancy not in complete remission.
2. Objectively confirmed catheter-related upper extremity DVT and treated with any standard therapeutic anticoagulation (including LMWH dose reduction to 75% after the first month) for at least 3 months.
3. Able and willing to provide informed consent.

Exclusion Criteria:

1. Active bleeding or other reasons for which anticoagulation is contraindicated.
2. Other indications requiring ongoing therapeutic dose of anticoagulation as deemed necessary by treating physicians (such as atrial fibrillation, mechanical heart valve, etc.).
3. Anticoagulation has been permanently stopped or reduced to prophylactic dose prior to enrollment for any reasons, except for participants who were transitioned to apixaban dosing regimen consistent with the protocol (2.5 mg twice daily) for ≤ 3 days .
4. Known contraindication for apixaban, such as allergy, hypersensitivity, or pregnancy.
5. Concomitant use of strong inhibitors or inducers of both cytochrome P450 3A4 (enzyme) and P-glycoprotein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Venous Thromboembolism (VTE) Rate | 6 months
  The rates of symptomatic, objectively confirmed new or recurrent major VTE (proximal upper or lower extremity DVT, segmental or larger pulmonary embolism (PE)) with corresponding 95% Confidence Interval (CI) at 6 months.

SECONDARY OUTCOMES:
Major Venous Thromboembolism (VTE) and Major bleeding Rate | 3 months
  Rates of new/recurrent symptomatic major VTE and major bleeding at 3 months.
New/recurrent symptomatic catheter-related upper extremity Deep Vein Thrombosis (DVT). | 3 months and 6 months
  New/recurrent symptomatic catheter-related upper extremity DVT.
New incidental Venous Thromboembolism (VTE) | 3 months and 6 months
  New incidental VTE (PE or upper or lower extremity DVT), defined as VTE diagnosed on imaging studies obtained not for concern of VTE, such as cancer staging scans.
New Deep Vein Thrombosis (DVT) | 3 months and 6 months
  New/recurrent any distal upper or lower extremity DVT or subsegmental PE.
Superficial vein thrombosis of upper or lower extremities | 3 months and 6 months
  Superficial vein thrombosis of upper or lower extremities
New unusual site Venous Thromboembolism (VTE) | 3 months and 6 months
  New unusual site VTE (such as splanchnic vein, cerebral vein, or gonadal vein thrombosis).
Clinically Relevant Non-Major Bleeding (CRNMB) events | 3 months and 6 months
  CRNMB events by International Society on Thrombosis and Haemostasis (ISTH) criteria2 and composite major bleeding and CRNMB events.
Arterial thromboembolic events | 3 months and 6 months
  Arterial thromboembolic events (objectively confirmed), including myocardial infarction, stroke, peripheral arterial disease, or other systemic arterial embolism.
All-cause mortality | 3 months and 6 months
  All-cause mortality
Correlative biomarkers | 6 months
  Correlative biomarkers at 6 months, while the exact list of correlative biomarkers is to be determined at the time of study completion, examples include D-dimer, P-selectin, prothrombin F1+F2, thrombin generation, etc.
Health-related quality of life using the EuroQoL-5D-5L Questionnaire | 6 months
  Health-related quality of life using EuroQoL-5D-5L (5Dimension- mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5L- severity levels) questionnaires on enrollment and at 6 months. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Fei Wang, MD, MPH, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No